CLINICAL TRIAL: NCT01840410
Title: A 12-month, Randomized, Double-masked, Sham-controlled, Multicenter Study to Evaluate the Efficacy and Safety of 0.5mg Ranibizumab Intravitreal Injections in Patients With Visual Impairment Due to Vascular Endothelial Growth Factor (VEGF) Driven Choroidal Neovascularization.
Brief Title: Assess the Efficacy/Safety of Intravitreal Ranibizumab in Patients With Vision Loss Due to Choroidal Neovascularization.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRFB002G2301; 2012-005417-38 (EudraCT Number)
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Choroidal Neovascularization (CNV)
Keywords: Vision Impairment; Abnormal growth of blood vessels
MeSH Terms: conditions — Choroidal Neovascularization; Vision Disorders | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab (Experimental): A 0.5 mg ranibizumab intravitreal injection was given to the study eye at baseline, and then as needed based on evidence of disease activity.
  Interventions: Drug: Ranibizumab
- Sham control (Sham Comparator): Sham injection was given to the study eye at baseline, and then treatment was given based on evidence of disease activity. At Month 1, if treatment was needed, sham was administered. At Month 2, participants could switch to open-label ranibizumab on an as needed basis.
  Interventions: Other: Sham control

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab 0.5mg/0.5mL was administered intravitreally to the participant.
  Arms: Ranibizumab
Other: Sham control — The sham vial did not contain active drug (empty sterile vial). The sham injection was an imitation of an intravitreal injection using an injection syringe without a needle touching the eye.
  Arms: Sham control

SUMMARY:
This study was conducted to evaluate the efficacy and safety of 0.5 mg ranibizumab in adult and adolescent patients with visual impairment due to choridal neovascularization (CNV).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of active CNV secondary to any causes with the CNV or its sequelae affecting the fovea;
* BCVA must be between ≥ 24 and ≤ 83 letters in the study eye;
* Visual loss in the study eye should mainly be due to the presence of any eligible types of CNV;

Key Exclusion Criteria:

* Women of child-bearing potential;
* Active malignancies;
* History of stroke less than 6 months prior to screening;
* Uncontrolled systemic inflammation or infection;
* Active diabetic retinopathy, active ocular/periocular infectious disease or active severe intra-ocular inflammation;
* CNV- conditions with a high likelihood of spontaneous resolution;
* History of intravitreal treatment with steroids;
* History of laser photocoagulation;
* History of intraocular treatment with any anti-angiogenic drugs.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (54):
- Australia (3):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, South Launceston, Tasmania
- Novartis Investigative Site, Montreal, Quebec, Canada
- Czechia (2):
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Glostrup Municipality, Denmark
- France (2):
  - Novartis Investigative Site, Paris, France
  - Novartis Investigative Site, Paris
- Germany (8):
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Regensburg, Germany
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Freiburg I. Br
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
- Greece (3):
  - Novartis Investigative Site, Pátrai, Greece
  - Novartis Investigative Site, Thessaloniki, Greece
  - Novartis Investigative Site, Heraklion Crete, GR
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Italy (6):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Varese, VA
- Novartis Investigative Site, Riga, Latvia
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Novartis Investigative Site, San Isidro, Lima region, Peru
- Poland (2):
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Wroclaw
- Portugal (2):
  - Novartis Investigative Site, Coimbra, Portugal
  - Novartis Investigative Site, Porto, Portugal
- Russia (2):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Banská Bystrica, Slovakia
  - Novartis Investigative Site, Trenčín, Slovakia
- South Korea (3):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seoul
- Spain (3):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Binningen
  - Novartis Investigative Site, Lausanne
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Kocaeli

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 183 participants were enrolled. Of these, 178 adults were randomized in a 2:1 ratio and considered for analysis. There were 5 adolescent participants, non-randomized, who received open-label treatment and were not included in the analyses. Therefore, the number enrolled = 183 differs from the participant flow number started = 178.
Period: Overall Study
Arm/Group | Ranibizumab | Sham Control
Started | 119 | 59
Safety Set | 119 | 59 (52 received ranibizumab at or after Month 2;7 did not receive ranibizumab any time during the study)
Full Analysis Set | 119 | 59
Completed | 112 | 55
Not Completed | 7 | 4
Not completed — Physician Decision | 1 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Protocol deviation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Sham Control | Total
Number analyzed (Participants) | 119 | 59 | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (15.07) | 51.9 (17.29) | 53.7 (15.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 30 | 90
  Male | 59 | 29 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) in Study Eye to Month 2
Description: BCVA was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity (VA) testing charts at an initial testing distance of 4 meters. The data were analyzed using mixed model repeated measures (MMRM) which contained scheduled visit, the type of underlying pathophysiologic mechanism (angloid streaks versus others) and treatment group as fixed effect factors, centered baseline BCVA as a continuous covariate and treatment group by visit and visit by centered baseline BCVA interactions. A positive change from baseline indicated improvement.
Time Frame: Baseline, Month 2
Population: The full analysis set (FAS) was considered for the analysis. The FAS included all participants who were randomized to treatment. Only participants, with available data at both baseline and Month 2, were analyzed.
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 118 | 57
letters | 9.5 (0.95) | -0.4 (1.16)
Statistical Analysis 1: Comparison: Ranibizumab vs Sham Control; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 9.94, 95% CI 2-sided [6.97 to 12.91], Standard Error of Mean 1.502

2. Secondary Outcome: Change From Baseline in BCVA in Study Eye up to Month 2
Description: BCVA was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity (VA) testing charts at an initial testing distance of 4 meters. The data were analyzed using analysis of covariance (ANCOVA) model which contained the type of underlying pathophysiologic mechanism (angloid streaks versus others) and treatment group as fixed effect factors, centered baseline BCVA as a continuous covariate. A positive change from baseline indicated improvement.
Time Frame: Baseline, Month 1, Month 2
Population: The full analysis set (FAS) was considered for the analysis. The FAS included all participants who were randomized to treatment. Only participants, with available data at both baseline and the given post-baseline time point, were analyzed for that post-baseline time point.
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 118 | 57
letters
  Month 1 | 7.1 (0.75) | 0.1 (1.08)
  Month 2 | 9.5 (0.91) | -0.4 (1.31)

3. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CSFT) in Study Eye
Description: CSFT was assessed by optical coherence tomography (OCT). A negative change from baseline indicates improvement.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometer (um)
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 119 | 59
micrometer (um)
  Month 1 (n=115,56) | -74.4 (81.25) | 3.3 (89.43)
  Month 2 (n=114,54) | -76.4 (108.24) | 1.9 (119.44)
  Month 3 (n=114,56) | -82.9 (114.26) | -59.1 (142.37)
  Month 4 (n=114,56) | -83.5 (104.71) | -68.4 (155.26)
  Month 5 (n=116,55) | -83.8 (112.41) | -89.4 (130.68)
  Month 6 (n=112,54) | -89.1 (109.19) | -85.9 (117.54)
  Month 7 (n=114,55) | -83.1 (105.97) | -84.5 (141.36)
  Month 8 (n=111,55) | -94.7 (111.54) | -97.9 (118.34)
  Month 9 (n=110,55) | -90.0 (112.44) | -93.5 (113.88)
  Month 10 (n=108,53) | -100.5 (119.45) | -85.4 (136.90)
  Month 11 (n=110,55) | -99.5 (112.38) | -82.8 (158.78)
  Month 12 (n=109,55) | -102.7 (117.27) | -91.7 (152.36)

4. Secondary Outcome: Change From Baseline in Central Subfield Volume (CSFV) in Study Eye
Description: CSFV was assessed OCT. A negative change from baseline indicates improvement.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microliter (ul)
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 119 | 59
microliter (ul)
  Month 1 (n=115,56) | -0.354 (0.4103) | 0.012 (0.3608)
  Month 2 (n=114,54) | -0.357 (0.5480) | -0.006 (0.5792)
  Month 3 (n=114,56) | -0.369 (0.5506) | -0.269 (0.6583)
  Month 4 (n=114,56) | -0.371 (0.4798) | -0.291 (0.7647)
  Month 5 (n=116,55) | -0.392 (0.5404) | -0.381 (0.5750)
  Month 6 (n=112,54) | -0.409 (0.5305) | -0.375 (0.5310)
  Month 7 (n=114,54) | -0.366 (0.4905) | -0.374 (0.5966)
  Month 8 (n=110,55) | -0.414 (0.5021) | -0.411 (0.4970)
  Month 9 (n=110,55) | -0.404 (0.5182) | -0.413 (0.5251)
  Month 10 (n=108,53) | -0.437 (0.5506) | -0.385 (0.5688)
  Month 11 (n=110,55) | -0.448 (0.5285) | -0.352 (0.7021)
  Month 12 (n=109,55) | -0.441 (0.5460) | -0.378 (0.6704)

5. Secondary Outcome: Number of Participants With Presence of Intra-retinal Fluid in Study Eye Compared to Baseline
Description: The presence of intra-retinal fluid was assessed by OCT.
Time Frame: Baseline, Month 2, Month 6, Month 12
Population: The FAS was considered for the analysis. The FAS included all randomized participants who received at least one dose of study treatment. Only participants (n), with values 'Absent' or 'Definite' for both the baseline and corresponding post-baseline time point, were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 119 | 59
Participants
  Baseline, Absent (n=116,56) | 70 | 32
  Baseline, Definite (n=116,56) | 46 | 24
  Month 2, Absent (n=116,56) | 97 | 29
  Month 2, Definite (n=116,56) | 19 | 27
  Month 6, Absent (n=116,54) | 100 | 43
  Month 6, Definite (n=116,54) | 16 | 11
  Month 12, Absent (n=111,55) | 95 | 45
  Month 12, Definite (n=111,55) | 16 | 10

6. Secondary Outcome: Number of Participants With Presence of Subretinal Fluid in Study Eye Compared to Baseline
Description: Presence of subretinal fluid in study eye compared to baseline
Time Frame: Baseline, Month 2, Month 6, Month 12
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 119 | 59
Participants
  Baseline, Absent (n=116,56) | 16 | 6
  Baseline, Definite (n=116,56) | 100 | 50
  Month 2, Absent (n=116,56) | 72 | 11
  Month 2, Definite (n=116,56) | 44 | 45
  Month 6, Absent (n=116,54) | 77 | 34
  Month 6, Definite (n=116,54) | 39 | 20
  Month 12, Absent (n=111,55) | 78 | 41
  Month 12, Definite (n=111,55) | 33 | 14

7. Secondary Outcome: Number of Participants With Presence of Active Chorioretinal Leakage
Description: The presence of active chorioretinal leakage was assessed by photography imaging, i.e. fluorescein angiography (FA).
Time Frame: Baseline, Month 2, Month 6, Month 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 119 | 59
Participants
  Baseline, Absent (n=106,50) | 2 | 1
  Baseline, Definite (n=106,50) | 104 | 49
  Month 2, Absent (n=106,50) | 37 | 4
  Month 2, Definite (n=106,50) | 69 | 46
  Month 6, Absent (n=108,45) | 64 | 29
  Month 6, Definite (n=108,45) | 44 | 16
  Month 12, Absent (n=103,47) | 81 | 37
  Month 12, Definite (n=103,47) | 22 | 10

8. Secondary Outcome: Average Change From Baseline in BCVA
Description: BCVA was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity (VA) testing charts at an initial testing distance of 4 meters. BCVA was assessed at each month from Month 1 through Month 6 or at each month from Month 1 through month 12, and the data were averaged. The outcome measure is reporting the change between baseline and average BCVA from Month 1 through Month 6 or from Month 1 through Month 12 (average BCVA - baseline BCVA). A positive change from baseline indicated improvement.
Time Frame: Baseline (BL), Month 1 through Month 6, Month 1 through Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 119 | 59
letters
  Average change from BL, month 1 through month 6 | 9.53 (10.467) | 4.68 (8.786)
  Average change from BL, month 1 through month 12 | 9.99 (11.528) | 6.59 (10.666)

9. Secondary Outcome: Number of Participants With ≥ 1, ≥ 5, ≥ 10 and ≥ 15 Letters Gain or Reaching 84 Letters
Description: VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using ETDRS-like visual acuity testing charts at a testing distance of 4 meters.
Time Frame: Month 2, Month 6, Month 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 119 | 59
Participants
  Month 2,>=15 letters or reaching 84 let.(n=118,57) | 37 | 7
  Month 2, >=10 letters (n=118,57) | 50 | 8
  Month 2, >=5 letters (n=118,57) | 83 | 16
  Month 2, >=1 letter (118,57) | 101 | 27
  Month 6,>=15 letters or reaching 84 let.(n=118,54) | 53 | 20
  Month 6, >=10 letters (n=118,54) | 67 | 24
  Month 6, >= 5 letters (n=118,54) | 88 | 34
  Month 6, >= 1 letter (n=118,54) | 104 | 39
  Month 12,>=15 letters or reaching 84 let.;n=113,55 | 55 | 23
  Month 12, >=10 letters (n=113,55) | 64 | 28
  Month 12, >=5 letters (n=113,55) | 81 | 34
  Month 12, >=1 letter (n=113,55) | 100 | 42

10. Secondary Outcome: Number of Participants With > 1, > 5, > 10 and > 15 Letters Loss
Description: as for outcome 9
Time Frame: Month 2, Month 6, Month 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 119 | 59
Participants
  Month 2, loss of >1 letter (n=118,57) | 10 | 24
  Month 2, loss of >5 letters (n=118,57) | 3 | 12
  Month 2, loss of >10 letters (n=118,57) | 1 | 5
  Month 2, loss of >15 letters (n=118,57) | 1 | 3
  Month 6, loss of >1 letter (n=118,54) | 10 | 9
  Month 6, loss of >5 letters (n=118,54) | 7 | 5
  Month 6, loss of >10 letters (n=118,54) | 6 | 2
  Month 6, loss of >15 letters (n=118,54) | 3 | 2
  Month 12, loss of >1 letter (n=113,55) | 9 | 10
  Month 12, loss of >5 letters (n=113,55) | 6 | 6
  Month 12, loss of >10 letters (n=113,55) | 5 | 4
  Month 12,loss of >15 letters (n=113,55) | 3 | 2

11. Secondary Outcome: Number of Participants With Requirement for Rescue Treatment at Month 1
Description: Rescue treatment with laser photocoagulation or periocular treatment could be administered at Month 1 only if the participant had a visual acuity loss of > 5 letters due to disease activity from baseline to Month 1.
Time Frame: Month 1
Population: The full analysis set (FAS) was considered for the analysis. The FAS included all participants who were randomized to treatment. Only participants, with available data at Month 1, were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Sham Control
Number analyzed (Participants) | 119 | 58
Participants | 0 | 1

12. Secondary Outcome: Number of Participants With Ranibizumab Treatments in Study Eye
Description: The number of participants administered study treatments, according to treatment frequency, was assessed.
Time Frame: Month 12
Population: Safety set: The safety set included randomized participants who received at least one dose of study treatment and was based on the actual treatment received.
Measure: Number; unit: Participants
Groups:
- Sham Without Ranibizumab: Participants did not receive ranibizumab at any time during the study.
Arm/Group | Ranibizumab | Sham Control | Sham Without Ranibizumab
Number analyzed (Participants) | 119 | 52 | 7
Participants
  Frequency of injections = 0 | 0 | 0 | 7
  Frequency of injections = 1 | 12 | 5 | 0
  Frequency of injections = 2 | 12 | 6 | 0
  Frequency of injections = 3 | 19 | 7 | 0
  Frequency of injections = 4 | 13 | 6 | 0
  Frequency of injections = 5 | 9 | 5 | 0
  Frequency of injections = 6 | 11 | 6 | 0
  Frequency of injections = 7 | 2 | 2 | 0
  Frequency of injections = 8 | 8 | 1 | 0
  Frequency of injections = 9 | 5 | 4 | 0
  Frequency of injections = 10 | 7 | 10 | 0
  Frequency of injections = 11 | 6 | 0 | 0
  Frequency of injections = 12 | 15 | 0 | 0

13. Secondary Outcome: Number of Participants With Re-treatments
Description: The number of participants, administered re-treatments according to treatment frequency, was assessed. Re-treatment was defined as an administration of study medication following at least one non-missed visit where treatment was not administered in the study eye. Up to month 12, the maximum number of retreatments was 5.
Time Frame: Month 12
Population: as for outcome 12
Measure: Number; unit: Paticipants
Arm/Group | Ranibizumab | Sham Control | Sham Without Ranibizumab
Number analyzed (Participants) | 119 | 52 | 7
Paticipants
  Frequency of re-treatment = 1 | 25 | 21 | 0
  Frequency of re-treatment = 2 | 22 | 10 | 0
  Frequency of re-treatment = 3 | 9 | 4 | 0
  Frequency of re-treatment = 4 | 5 | 2 | 0

14. Secondary Outcome: Number of Primary Reasons for Decision to Treat by Investigator
Description: The total number of primary reasons for decisions to treat was assessed. A single participant could have had multiple primary reasons for treatment.
Time Frame: Month 12
Population: as for outcome 12
Measure: Number; unit: Number of primary reasons
Units Other Than Participants: treatment decisions
Arm/Group | Ranibizumab | Sham Control | Sham Without Ranibizumab
Number analyzed (Participants) | 119 | 52 | 7
Number analyzed (treatment decisions) | 580 | 328 | 1
Number of primary reasons
  Vision impairment | 29 | 9 | 0
  OCT abnormality | 522 | 306 | 1
  FA abnormality | 21 | 13 | 0
  Color fundus photography abnormality | 1 | 0 | 0
  Clinical abnormality | 6 | 0 | 0
  Without documentation | 1 | 0 | 0

ADVERSE EVENTS:
Groups:
- Sham With Ranibizumab: Sham injection was given to the study eye at baseline, and then treatment was given based on evidence of disease activity. At month 1, if treatment was needed, sham was administered. At month 2, participants switched to open-label ranibizumab on an as needed basis.
Arm/Group | Ranibizumab | Sham With Ranibizumab | Sham Without Ranibizumab
Serious Adverse Events (participants affected / at risk) | 9/119 | 4/52 | 0/7
Other Adverse Events (participants affected / at risk) | 42/119 | 19/52 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=119) | Sham With Ranibizumab (N=52) | Sham Without Ranibizumab (N=7)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Retinal detachment (Fellow untreated eye) (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=119) | Sham With Ranibizumab (N=52) | Sham Without Ranibizumab (N=7)
Choroidal neovascularisation (Study eye) (Eye disorders) | 3 | 0 | 1
Conjunctival haemorrhage (Study eye) (Eye disorders) | 7 | 6 | 0
Eye inflammation (Study eye) (Eye disorders) | 0 | 0 | 1
Foreign body sensation in eyes (Study eye) (Eye disorders) | 1 | 1 | 1
Macular oedema (Study eye) (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Study eye) (Eye disorders) | 1 | 1 | 1
Photopsia (Study eye) (Eye disorders) | 1 | 0 | 1
Visual acuity reduced (Study eye) (Eye disorders) | 3 | 1 | 1
Conjunctivitis (Study eye) (Infections and infestations) | 2 | 3 | 0
Influenza (Infections and infestations) | 9 | 0 | 0
Nasopharyngitis (Infections and infestations) | 14 | 9 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1
Headache (Nervous system disorders) | 1 | 3 | 1
Hypertension (Vascular disorders) | 5 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.